CLINICAL TRIAL: NCT00425984
Title: Randomized Trial of Male Circumcision for HIV Prevention, Rakai, Uganda
Brief Title: Male Circumcision for HIV Prevention in Rakai, Uganda
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U1AI171-1-02; U1 AII 171-01-02; U1 AI 171-1-02
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2007-08-24 (Estimated); Status verified 2007-08

CONDITIONS: HIV Infections; Herpesvirus 2, Human; Syphilis; Genital Diseases, Male
Keywords: HIV; Male circumcision; Sexually transmitted infections; Sexual risk behaviors; Adult males; Haemophilus ducreyi; Human papillomavirus; Rakai; Uganda; HIV seronegativity; HPV; STI
MeSH Terms: conditions — HIV Infections; Syphilis; Genital Diseases, Male; Sexually Transmitted Diseases; Chancroid

INTERVENTIONS:
Procedure: Adult male circumcision

SUMMARY:
Circumcision in HIV unifected men may reduce the likelihood of becoming infected with HIV, reduce sexually transmitted infections (STIs) in men, not engender increases in sexual risk behaviors, and be acceptable to men as a procedure for preventing HIV. The purpose of this study is to evaluate circumcision in HIV uninfected men in terms of safety and ability to prevent HIV infection.

DETAILED DESCRIPTION:
South Africa has one of the most severe and fast-growing HIV epidemics in the world. Adult male circumcision may be an effective preventive measure to slow the spread of HIV and other STIs. This study will assess the efficacy of circumcision in HIV uninfected men in preventing HIV and STI acquisition.

This study will have two stages. In the first stage, 200 men will be enrolled into a study of the acceptability, feasibility, and safety of circumcision. Frequent postoperative follow-up will occur to determine rates of healing and complications. After assessment of those enrolled in Stage 1, Stage 2 enrollment will begin. Stage 2 will determine the efficacy of circumcision in preventing HIV acquisition. In both stages, HIV uninfected men will be randomly assigned to have either immediate circumcision or possible circumcision 2 years following Stage 2 study entry. The participants not receiving immediate circumcision will be offered circumcision after completion of 2 years of follow-up study, provided there is evidence of the efficacy of this procedure at that time. If efficacy is still unknown after 2 years of follow-up, participants will be given the option of circumcision at the completion of the trial.

Postoperative follow-up visits will be scheduled between 24 to 48 hours, 5 to 9 days, and 4 to 6 weeks. At each postoperative visit, participants will be questioned about symptoms suggestive of complications, and the area operated on will be inspected. Participants will be asked about resumption of sexual intercourse, and those who have resumed sexual intercourse will be asked about condom use. Study visits will be also conducted regarding risk behaviors and symptoms of STIs, and these will occur sometime between Weeks 4 to 6, and at Months 6, 12, and 24 post-enrollment. At each study visit, assessment of circumcision status and penile pathology; blood, urine, and penile swabs collection; and HIV testing will occur, and counseling and health education will be provided.

ELIGIBILITY:
Inclusion Criteria:

* HIV uninfected
* Willing to receive HIV results
* Willing to be circumcised
* Parent or guardian willing to provide informed consent if applicable
* Hemoglobin of 8 grams/dl or less
* Intend to stay in Rakai, Uganda, for at least 1 year and are available for follow-up for 1 year

Exclusion Criteria:

* Already circumcised or partially circumcised
* Anatomical abnormality of the penis (e.g., hypospadias, severe phimosis) that may put the participant at risk if circumcised
* Medical conditions that require therapeutic circumcision
* Medical condition that contraindicates surgery or use of local anesthesia

Ages: 15 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5000
Dates: Start 2002-08; Study Completion 2006-12

PRIMARY OUTCOMES:
HIV acquisition
safety of circumcision

SECONDARY OUTCOMES:
Sexually transmitted infections
sexual risk behaviors
acceptability

CONTACTS AND LOCATIONS:
Overall Officials: Ronald H. Gray, MD, Principal Investigator — Department of Population, Family and Reproductive Health Sciences, Bloomberg School of Public Health, Johns Hopkins University
Locations (1):
- Rakai Health Sciences Program, P.O. Box 279, Kalisizo Town, Rakai, Uganda

REFERENCES:
- [Background] de Bruyn G, Smith MD, Gray GE, McIntyre JA, Wesson R, Dos Passos G, Martinson NA. Circumcision for prevention against HIV: marked seasonal variation in demand and potential public sector readiness in Soweto, South Africa. Implement Sci. 2007 Jan 25;2:2. doi: 10.1186/1748-5908-2-2. PMID 17254337
- [Background] Gray RH, Kiwanuka N, Quinn TC, Sewankambo NK, Serwadda D, Mangen FW, Lutalo T, Nalugoda F, Kelly R, Meehan M, Chen MZ, Li C, Wawer MJ. Male circumcision and HIV acquisition and transmission: cohort studies in Rakai, Uganda. Rakai Project Team. AIDS. 2000 Oct 20;14(15):2371-81. doi: 10.1097/00002030-200010200-00019. PMID 11089626
- [Background] Kelly R, Kiwanuka N, Wawer MJ, Serwadda D, Sewankambo NK, Wabwire-Mangen F, Li C, Konde-Lule JK, Lutalo T, Makumbi F, Gray RH. Age of male circumcision and risk of prevalent HIV infection in rural Uganda. AIDS. 1999 Feb 25;13(3):399-405. doi: 10.1097/00002030-199902250-00013. PMID 10199231
- [Background] Wawer MJ, Reynolds SJ, Serwadda D, Kigozi G, Kiwanuka N, Gray RH. Might male circumcision be more protective against HIV in the highly exposed? An immunological hypothesis. AIDS. 2005 Dec 2;19(18):2181-2. doi: 10.1097/01.aids.0000194132.51006.4f. No abstract available. PMID 16284475
- [Result] Gray RH, Kigozi G, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chaudhary MA, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Williams CF, Opendi P, Reynolds SJ, Laeyendecker O, Quinn TC, Wawer MJ. Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial. Lancet. 2007 Feb 24;369(9562):657-66. doi: 10.1016/S0140-6736(07)60313-4. PMID 17321311
- [Derived] Grabowski MK, Gray RH, Makumbi F, Kagaayi J, Redd AD, Kigozi G, Reynolds SJ, Nalugoda F, Lutalo T, Wawer MJ, Serwadda D, Quinn TC, Tobian AAR. Use of injectable hormonal contraception and women's risk of herpes simplex virus type 2 acquisition: a prospective study of couples in Rakai, Uganda. Lancet Glob Health. 2015 Aug;3(8):e478-e486. doi: 10.1016/S2214-109X(15)00086-8. Epub 2015 Jun 17. PMID 26094162
- [Derived] Gray R, Kigozi G, Kong X, Ssempiija V, Makumbi F, Wattya S, Serwadda D, Nalugoda F, Sewenkambo NK, Wawer MJ. The effectiveness of male circumcision for HIV prevention and effects on risk behaviors in a posttrial follow-up study. AIDS. 2012 Mar 13;26(5):609-15. doi: 10.1097/QAD.0b013e3283504a3f. PMID 22210632
- [Derived] Wawer MJ, Tobian AA, Kigozi G, Kong X, Gravitt PE, Serwadda D, Nalugoda F, Makumbi F, Ssempiija V, Sewankambo N, Watya S, Eaton KP, Oliver AE, Chen MZ, Reynolds SJ, Quinn TC, Gray RH. Effect of circumcision of HIV-negative men on transmission of human papillomavirus to HIV-negative women: a randomised trial in Rakai, Uganda. Lancet. 2011 Jan 15;377(9761):209-18. doi: 10.1016/S0140-6736(10)61967-8. Epub 2011 Jan 6. PMID 21216000
- [Derived] Gray RH, Serwadda D, Kong X, Makumbi F, Kigozi G, Gravitt PE, Watya S, Nalugoda F, Ssempijja V, Tobian AA, Kiwanuka N, Moulton LH, Sewankambo NK, Reynolds SJ, Quinn TC, Iga B, Laeyendecker O, Oliver AE, Wawer MJ. Male circumcision decreases acquisition and increases clearance of high-risk human papillomavirus in HIV-negative men: a randomized trial in Rakai, Uganda. J Infect Dis. 2010 May 15;201(10):1455-62. doi: 10.1086/652184. PMID 20370483
- [Derived] Gray RH, Serwadda D, Tobian AA, Chen MZ, Makumbi F, Suntoke T, Kigozi G, Nalugoda F, Iga B, Quinn TC, Moulton LH, Laeyendecker O, Reynolds SJ, Kong X, Wawer MJ. Effects of genital ulcer disease and herpes simplex virus type 2 on the efficacy of male circumcision for HIV prevention: Analyses from the Rakai trials. PLoS Med. 2009 Nov;6(11):e1000187. doi: 10.1371/journal.pmed.1000187. Epub 2009 Nov 24. PMID 19936044
- [Derived] Mehta SD, Gray RH, Auvert B, Moses S, Kigozi G, Taljaard D, Puren A, Agot K, Serwadda D, Parker CB, Wawer MJ, Bailey RC. Does sex in the early period after circumcision increase HIV-seroconversion risk? Pooled analysis of adult male circumcision clinical trials. AIDS. 2009 Jul 31;23(12):1557-64. doi: 10.1097/QAD.0b013e32832afe95. PMID 19571722
- [Derived] Kiggundu V, Watya S, Kigozi G, Serwadda D, Nalugoda F, Buwembo D, Settuba A, Anyokorit M, Nkale J, Kighoma N, Ssempijja V, Wawer M, Gray RH. The number of procedures required to achieve optimal competency with male circumcision: findings from a randomized trial in Rakai, Uganda. BJU Int. 2009 Aug;104(4):529-32. doi: 10.1111/j.1464-410X.2009.08420.x. Epub 2009 Apr 21. PMID 19389002
- [Derived] Tobian AA, Serwadda D, Quinn TC, Kigozi G, Gravitt PE, Laeyendecker O, Charvat B, Ssempijja V, Riedesel M, Oliver AE, Nowak RG, Moulton LH, Chen MZ, Reynolds SJ, Wawer MJ, Gray RH. Male circumcision for the prevention of HSV-2 and HPV infections and syphilis. N Engl J Med. 2009 Mar 26;360(13):1298-309. doi: 10.1056/NEJMoa0802556. PMID 19321868
- [Derived] Tobian AA, Charvat B, Ssempijja V, Kigozi G, Serwadda D, Makumbi F, Iga B, Laeyendecker O, Riedesel M, Oliver A, Chen MZ, Reynolds SJ, Wawer MJ, Gray RH, Quinn TC. Factors associated with the prevalence and incidence of herpes simplex virus type 2 infection among men in Rakai, Uganda. J Infect Dis. 2009 Apr 1;199(7):945-9. doi: 10.1086/597074. PMID 19220138
- [Derived] Kigozi G, Gray RH, Wawer MJ, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Ridzon R, Opendi P, Sempijja V, Settuba A, Buwembo D, Kiggundu V, Anyokorit M, Nkale J, Kighoma N, Charvat B. The safety of adult male circumcision in HIV-infected and uninfected men in Rakai, Uganda. PLoS Med. 2008 Jun 3;5(6):e116. doi: 10.1371/journal.pmed.0050116. PMID 18532873
- [Derived] Kigozi G, Watya S, Polis CB, Buwembo D, Kiggundu V, Wawer MJ, Serwadda D, Nalugoda F, Kiwanuka N, Bacon MC, Ssempijja V, Makumbi F, Gray RH. The effect of male circumcision on sexual satisfaction and function, results from a randomized trial of male circumcision for human immunodeficiency virus prevention, Rakai, Uganda. BJU Int. 2008 Jan;101(1):65-70. doi: 10.1111/j.1464-410X.2007.07369.x. PMID 18086100
- [Derived] Gray RH, Makumbi F, Serwadda D, Lutalo T, Nalugoda F, Opendi P, Kigozi G, Reynolds SJ, Sewankambo NK, Wawer MJ. Limitations of rapid HIV-1 tests during screening for trials in Uganda: diagnostic test accuracy study. BMJ. 2007 Jul 28;335(7612):188. doi: 10.1136/bmj.39210.582801.BE. Epub 2007 Jun 1. PMID 17545184